CLINICAL TRIAL: NCT00710463
Title: Evaluation of the Role of Nocturnal Non-Invasive Ventilation in Pulmonary Rehabilitation
Status: Completed | Type: Observational
Sponsor: Deutsche Lungenstiftung e.V. (Other)
Collaborators: Hannover Medical School (Other)
Responsible Party: Dr. Klaus Kenn, Klinikum Berchtesgadener Land, Malterhöh 1, D-83471 Berchtesgaden
Other Study IDs: NIV and Rehabilitation
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; non invasive ventilation; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: patients receive a hospital based comprehensive pulmonary rehabilitation programme, including endurance training, physiotherapy, medical therapy, and long term oxygen treatment when indicated.
- NIV treatment group: patients receive a hospital based comprehensive pulmonary rehabilitation programme, including endurance training, physiotherapy, medical therapy, and long term oxygen treatment when indicated, plus newly introduced nocturnal non invasive ventilation.
  Interventions: Device: non invasive ventilation (Resmed VPAP III ST-A, Respironics Harmony)

INTERVENTIONS:
Device: non invasive ventilation (Resmed VPAP III ST-A, Respironics Harmony) — non invasive ventilation was performed with commercially available ventilators from the manufacturers Resmed and Respironics.
  Other Names: Resmed VPAP III ST-A; Respironics Harmony
  Groups: NIV treatment group

SUMMARY:
Hypothesis: Hospital based, comprehensive pulmonary rehabilitation of patients with COPD in GOLD stage IV can be optimized by application of nocturnal non invasive ventilation.

This hypotheses shall be tested by an observational trial, comparing rehabilitation effects of a prospectively observed group receiving non invasive ventilation, compared wiht a historical control group of patients who did received the same treatment without non invasive ventilation.

DETAILED DESCRIPTION:
Non invasive ventilation is known to allow improvements if applied during endurance training, but this is technically difficult. Nocturnal application of non invasive ventilation is known to unload the ventilatory pump, reset the control of breathing, and improve sleep quality.

The protocol also aimed to evaluate the acceptance of non invasive ventilation in patients undergoing a four week inpatient pulmonary rehabilitation programme.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COPD in stages GOLD IV
* Receiving optimized medical treatment and long term oxygen treatment, if indicated
* Patient's consent to participate in this trial

Exclusion Criteria:

* Previous treatment with NIPPV
* Unwillingness or intolerance to perform NIPPV
* Acute exacerbation of COPD at baseline or during pulmonary rehabilitation,
* Significant orthopaedic or neurologic problems that reduce mobility or cooperation with physical training
* Poor controlled coexisting psychiatric or unstable cardiac disease,
* Inability to perform a six minute walk test
* Extreme hypercapnia (pCO2 > 74 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients were recruited at a single center, the rehabilitation hospital "Klinikum Berchtesgadener Land" at Germany.
  Patients entering the well defined, hospital based pulmonary rehabilitation programme after Januar 1, 2005 were additionally treated with nocturnal non invasive ventilation. The results of these patients were compared with a group of patients who underwent the same rehabilitation programme in the years 2003 to 2005, when non invasive ventilation was not availabe.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2003-05; Primary Completion 2007-09 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
six minute walk distance | beginning to end of rehabilitation

SECONDARY OUTCOMES:
quality of life | beginning to end of rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, MD, Study Director — Klinikum Berchtesgadener Land; Ursula Schönheit-Kenn, ME, Principal Investigator — Klinikum Berchtesgadener Land
Locations (1):
- Klinikum Berchtesgadener Land, Berchtesgaden, Germany